CLINICAL TRIAL: NCT05445388
Title: Feasibility of Structural and Functional Imaging of the Middle Ear and Its Constituents by Optical Coherence Tomography
Brief Title: Feasibility of Middle Ear OCT Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. R.M. Metselaar MD, PhD, Dr. R.M. Metselaar MD PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL81519.078.22
Record Dates: First submitted 2022-06-17; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Image, Body
Keywords: Middle Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT imaging (Experimental): OCT imaging
  Interventions: Device: Aurisvue

INTERVENTIONS:
Device: Aurisvue — OCT imaging of the middle ear

SUMMARY:
Feasibility of structural and functional imaging of the middle ear and its constituents by optical coherence tomography.

DETAILED DESCRIPTION:
Rationale: Various middle ear diseases can affect anatomical structures of the middle ear in different ways. Unfortunately, current methods for assessing the structure and function of the constituents of the middle ear are limited and often fail to provide all clinically relevant data. Optical coherence tomography (OCT) is a technology that can provide valuable, additional information with a newly developed prototype OCT-device for structural and functional imaging of the middle ear.

Objective: To assess the feasibility and the clinical potential of structural and functional OCT imaging with a newly developed OCT-device in patients with various middle ear problems.

Study design: Observational study Study population: Adult patients presenting with various middle ear complaints at the Ear Nose Throat department of the Department of Otorhinolaryngology and Head and Neck Surgery, Erasmus Medical Center, Rotterdam, the Netherlands.

Main study parameters/endpoints: Percentage of patients in which structural OCT imaging was feasible (i.e., the OCT images showed a discernible tympanic membrane (TM) and at least one of the ossicles).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden is minimal: patient examination with Aurisvue is similar to the conventional examination with a standard otoscope and will take approximately 5 to 10 minutes. The risks are negligible: imaging is done with light levels well below the maximum permissible exposure level and sound levels to induce movement of the TM and the ossicular chain are well below the hazardous threshold.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* competent, willing and able to cooperate

Exclusion Criteria:

* any acute or chronic condition that would limit the ability of the patient to participate in the study, per attending physician's indication
* refusal to give informed consent
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Middle ear structures identified with the Aurisvue OCT device | 1 Year
  Identification of each of the following anatomical middle ear structures with Aurisvue: tympanic membrane, malleus, incus, stapes and promontory (visible or not visible)

SECONDARY OUTCOMES:
OCT-vibrometry measurements with the Aurisvue OCT device | 1 Year
  Number of middle ear structures (tympanic membrane, malleus, incus and stapes) on which OCT-vibrometry measurements by Aurisvue succeeded.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT05445388/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT05445388/ICF_001.pdf